CLINICAL TRIAL: NCT01598844
Title: The JenaValve" EvalUation of Long Term Performance and Safety In PaTients With SEvere Aortic Stenosis oR Aortic Insufficiency
Brief Title: JUPITER Study: Transapical Aortic Valve Implantation for Aortic Regurgitation
Acronym: JUPITER
Status: Completed | Type: Observational
Sponsor: JenaValve Technology, Inc. (Industry)
Collaborators: King's College London (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: JV03PMS
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Aortic Stenosis; Aortic Insufficiency; Aortic Regurgitation
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High risk patients with aortic stenosis: Transapical aortic valve implantation using a transcatheter heart valve for aortic stenosis.
  Interventions: Device: Transcatheter aortic valve replacement
- High risk patients with AI: Transapical aortic valve implantation using a transcatheter heart valve for aortic regurgitation.
  Interventions: Device: Transcatheter aortic valve replacement

INTERVENTIONS:
Device: Transcatheter aortic valve replacement — Transcatheter aortic valve replacement via a transapical access
  Other Names: The JenaValve TAVI System

SUMMARY:
The purpose of this registry is to observe longterm performance and safety of the JenaValve TAVI system, in routine medical and everyday conditions.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the long term safety and effectiveness of the CE-marked JenaValve System Transapical in an elderly patient population with severe aortic stenosis and/or aortic insufficiency who are at high risk for open surgical aortic valve replacement.

The target study population will consist of elderly patients suffering from severe symptomatic degenerative aortic valve stenosis and/or aortic insufficiency who show an increased risk for an open aortic valve replacement surgery due to existing co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for TAVI with the JenaValve according to instructions for use

Exclusion Criteria:

* Patients unsuitable for TAVI with the JenaValve according to instructions for use

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe aortic stenosis or with severe aortic insufficiency and an increased risk for an open aortic valve replacement surgery
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2012-05-30 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 day
  30-day mortality of procedure is defined as all deaths within 30 days after implantation of the JenaValve prosthesis irrespective of the underlying cause of death.

SECONDARY OUTCOMES:
Safety Endpoints | peri- and post-operatively and at 3, 6, 12, 24 and 36 months
  * All-cause mortality
  * Cardiovascular mortality
  * Major stroke
  * Life-threatening or disabling bleeding
  * Major bleeding
  * Acute kidney injury
  * Myocardial infarction
  * Major vascular complication
  * Mechanical coronary obstruction
  * Prosthetic valve thrombus
  * Prosthetic valve endocarditis
  * Conduction disturbance and cardiac arrhythmia
  * Necessity of permanent pacemaker implantation
Device Success | Index Procedure and Immediate Post-operative
  The following parameters will be collected to assess device success:
  1. Successful vascular access, delivery and deployment of the device successful retrieval of the device
  2. Correct position of the device in the proper anatomical location
  3. Intended performance of the prosthetic heart valve:
  4. Only one valve implanted in proper anatomical position
Device Effectiveness | Prior to discharge, at 3, 6, 12, 24 and 36 months
  The following parameters will assess effectiveness:
  * Transvalvular aortic peak pressure gradient
  * Transvalvular aortic mean pressure gradient
  * Effective aortic valve area
  * Paravalvular regurgitation coded according to VARC
  * Transvalvular regurgitation coded according to VARC
  * No clinically significant valve migration/dislocation
  * Absence of mechanical coronary obstruction
  * Functional improvement assessment by NYHA functional classification
SF-12 Survey of Quality of Life | at 12 months
  The SF-12 health survey to measure mental and physical health of the patient.
Combined Safety Endpoint | at 30 days
  A combined safety endpoint will be assessed at 30 days consisting of the following variables:
  * All-cause mortality
  * Major stroke
  * Acute kidney injury (Stage 3)
  * Life-threatening or disabling bleeding
  * Major vascular complication
  * Peri-procedural myocardial infarction
  * Repeat surgical or interventional procedure for valve-related dysfunction
Combined Efficacy Endpoint | at 12 months
  A combined efficacy endpoint will be assessed consisting of the following variables:
  * All-cause mortality (after > 30 days)
  * Failure of current therapy for AS, requiring hospitalization for symptoms of valve-related or cardiac decompensation
  * Prosthetic heart valve dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Wendler, Prof, Principal Investigator — King's College Hospital NHS Trust; Hendrik Treede, Prof, Principal Investigator — University Heart Center Hamburg
Locations (15):
- Germany (12):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Herzzentrum der Universität, Cologne
  - Herzzentrum Dresden, Universitätsklinik an der Technischen Universität Dresden, Dresden
  - University Hospital, Erlangen
  - University Heart Centre, Freiburg im Breisgau
  - Asklepios Klinik, Hamburg
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Herzzentrum Leipzig - Universitätsklinik, Leipzig
  - Deutsches Herzzentrum München, Munich
  - Herzzentrum des Städtischen Klinikums München, Munich
  - Herz- und Kreislaufzentrum Rotenburg (Fulda), Rotenburg an der Fulda
  - Robert Bosch Krankenhaus Stuttgart, Stuttgart
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Universitätsspital Basel, Basel, Switzerland
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Background] Mieres J, Menendez M, Fernandez-Pereira C, Rubio M, Rodriguez AE. Transapical Implantation of a 2nd-Generation JenaValve Device in Patient with Extremely High Surgical Risk. Case Rep Cardiol. 2015;2015:458151. doi: 10.1155/2015/458151. Epub 2015 Aug 4. PMID 26346128
- [Background] Seiffert M, Bader R, Kappert U, Rastan A, Krapf S, Bleiziffer S, Hofmann S, Arnold M, Kallenbach K, Conradi L, Schlingloff F, Wilbring M, Schafer U, Diemert P, Treede H. Initial German experience with transapical implantation of a second-generation transcatheter heart valve for the treatment of aortic regurgitation. JACC Cardiovasc Interv. 2014 Oct;7(10):1168-74. doi: 10.1016/j.jcin.2014.05.014. Epub 2014 Aug 13. PMID 25129672
- [Result] Silaschi M, Treede H, Rastan AJ, Baumbach H, Beyersdorf F, Kappert U, Eichinger W, Ruter F, de Kroon TL, Lange R, Ensminger S, Wendler O. The JUPITER registry: 1-year results of transapical aortic valve implantation using a second-generation transcatheter heart valve in patients with aortic stenosis. Eur J Cardiothorac Surg. 2016 Nov;50(5):874-881. doi: 10.1093/ejcts/ezw170. Epub 2016 May 30. PMID 27242354
- [Result] Silaschi M, Conradi L, Wendler O, Schlingloff F, Kappert U, Rastan AJ, Baumbach H, Holzhey D, Eichinger W, Bader R, Treede H. The JUPITER registry: One-year outcomes of transapical aortic valve implantation using a second generation transcatheter heart valve for aortic regurgitation. Catheter Cardiovasc Interv. 2018 Jun;91(7):1345-1351. doi: 10.1002/ccd.27370. Epub 2017 Nov 24. PMID 29171730